CLINICAL TRIAL: NCT04763057
Title: Calcium Hydroxide Versus NeoPUTTY MTA in Indirect Pulp Treatment of Primary Molars: A Randomized Clinical Trial
Brief Title: Indirect Pulp Treatment in Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa aly fouad elchaghaby, Lecturer of Pediatric Dentistry and Dental public health, Faculty of Dentistry, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vital pulp treatment
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Deep Caries
MeSH Terms: interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indirect pulp treatment with NeoPUTTY MTA (Experimental)
  Interventions: Drug: NeoPUTTY MTA
- indirect pulp treatment with calcium hydroxide (Active Comparator)
  Interventions: Drug: calcium hydroxide

INTERVENTIONS:
Drug: NeoPUTTY MTA — NeoPUTTY, a premixed bioactive bioceramic MTA that triggers hydroxyapatite and supports healing
  Arms: indirect pulp treatment with NeoPUTTY MTA
Drug: calcium hydroxide — Calcium hydroxide the gold standard for IPT
  Arms: indirect pulp treatment with calcium hydroxide

SUMMARY:
Conservative approaches such as indirect pulp capping techniques became popular over the last years for the management of deep carious lesions. In particular, indirect pulp-treatment (IPT) techniques have gained remarkable attention in pediatric dentistry, mainly because children require a fast and accurate treatment, besides it enables the affected primary tooth to remain in the mouth until exfoliation without causing any pain or infection.

DETAILED DESCRIPTION:
Indirect pulp treatment is recommended for teeth with deep caries approximating the pulp with no signs and symptoms of pulp deterioration. In this treatment, the deepest layer of the remaining carious dentine (affected dentin) is covered with biocompatible material followed by an airtight restoration to achieve a good seal against microleakage, without the need to reencounter for the removal of remaining caries.

Calcium hydroxide has served as a gold standard for IPT over the years. However, the introduction of newer bioactive materials such as mineral trioxide aggregate (MTA) and Biodentine helped surpass the demerits of calcium hydroxide such as internal resorption, nonadherence to dentin, degradation over time, tunnel defects, and poor sealing ability.

ELIGIBILITY:
Inclusion Criteria:

* • Presence of active carious lesions involving either occlusal or proximal surfaces of primary molars.

  * Extension of carious lesion such that complete caries removal would risk pulp exposure.
  * History of tolerable dull intermittent pain, mild discomfort associated with eating, negative history of spontaneous extreme pain.
  * Radiographically, carious lesion involving more than 2/3rd thickness of dentin approximating the pulp, normal lamina dura, normal periodontal ligament space, more than 2/3rd of root present, no periapical changes, no pathologic external or internal resorption.

Exclusion Criteria:

* • History of spontaneous sharp, penetrating pain, or tenderness on percussion

  * Presence of tooth mobility, discoloration, sinus opening, or abscessed tooth.
  * Radiographically, presence of interrupted or broken lamina dura, widened periodontal ligament space, periapical radiolucency, internal or external resorption.
  * Pulp exposure during caries removal.
  * Parental refusal for participation.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success in term of the absence of post-operative pain | one year
  Visual analog scale
Clinical success in term of the absence of pain on percussion, swelling, sinus, or fistula | one year
  Visual and clinical examinations

SECONDARY OUTCOMES:
Radiographic success in term of the absence of any adverse radiographic findings (eg. internal or external root resorption or other pathologic changes | one year
  Radiographic examination